CLINICAL TRIAL: NCT01589588
Title: Administration of Oxygen to Cluster Headache Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mads Barløse (Other)
Responsible Party: Sponsor-Investigator, Mads Barløse, MD, principal investigator, Danish Headache Center
Organization: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-2-2011-163
Record Dates: First submitted 2012-04-26; First posted 2012-05-02 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Cluster Headache Attacks
Keywords: acute treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (4):
- Mask 1 (Experimental)
  Interventions: Device: Open Hudson Mask
- Mask 2 (Experimental)
  Interventions: Device: Cluster headache mask with 3 L reservoir
- Mask 3 (Experimental)
  Interventions: Device: Mask 3; Device: Carnét oxygen demand valve
- Mask 3, placebo (Placebo Comparator)
  Interventions: Device: Carnét oxygen demand valve

INTERVENTIONS:
Device: Open Hudson Mask — Mask type 1 oxygen
  Arms: Mask 1
Device: Cluster headache mask with 3 L reservoir — Mask type 2 with oxygen
  Arms: Mask 2
Device: Mask 3 — Mask type 3 oxygen
  Arms: Mask 3
Device: Carnét oxygen demand valve — mask type 3 oxygen
  Arms: Mask 3
Device: Carnét oxygen demand valve — mask type 3 placebo
  Arms: Mask 3, placebo

SUMMARY:
This study will investigate the possible difference in treatment effect between three different oxygen delivery systems in the acute treatment of cluster headaches.

ELIGIBILITY:
Inclusion Criteria:

* episodic cluster headache
* regular occurance of attacks and cluster for 2 years
* 2-8 attacks / day
* cluster periods of over 14 days
* duration of current cluster period max 14 days
* ability to differentiate between attacks of CH and other forms of headache

Exclusion Criteria:

* Changes in prophylactic treatment a week before trial
* pregnancy or breastfeeding women
* serious somatic or psychiatric disease
* COLD
* chronic or primary or secondary headache > 14 days / month other than CH
* alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 15 minutes
  Pain relief after 15 minutes of treatment

SECONDARY OUTCOMES:
Mask preference | 2 days
  subject mask preference

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark